CLINICAL TRIAL: NCT06199180
Title: Pulsed Field Ablation Versus Conventional Radiofrequency Catheter Ablation for Repeat
Brief Title: Pulsed Field Ablation Versus Conventional Radiofrequency Catheter Ablation for Repeat PVI in Patients With Paroxysmal AF
Acronym: REPEAT-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REPEAT-AF trial
Record Dates: First submitted 2023-12-01; First posted 2024-01-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation Recurrent
Keywords: pulmonary vein isolation; pulsed field ablation; radiofrequency ablation; implantable cardiac monitor
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: patients will be randomised to PFA or RFA for redo PVI
Who Masked: Outcomes Assessor
Masking Description: Patients know their treatment arm. All endpoints will be adjudicated by a blinded endpoint committee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation (Active Comparator): In this group, patients will undergo the acquisition of a 3D high-density map. If pulmonary vein (PV) reconnection is identified, radiofrequency ablation (RFA) will be employed for pulmonary vein isolation (PVI). Should PV reconnection not be detected, the operator will have the discretion to determine the necessary ablation strategies. Patients falling into this category will be included in a concurrent registry.
  Interventions: Device: pulmonary vein isolation with RFA
- Pulsed field ablation (Experimental): In this group, pulmonary vein (PV) reconnection is identified by the FARAWAVE system. If reconnection is observed, pulsed field ablation (PFA) will be employed for pulmonary vein isolation (PVI). Should PV reconnection not be detected, the operator will have the discretion to determine the necessary ablation strategies. Patients falling into this category will be included in a concurrent registry.
  Interventions: Device: pulmonary vein isolation with PFA

INTERVENTIONS:
Device: pulmonary vein isolation with RFA — Patients randomised to RFA will undergo PVI with point-by-point RFA.
  Arms: Radiofrequency ablation
Device: pulmonary vein isolation with PFA — Patients randomised to PFA will undergo PVI with PFA.
  Arms: Pulsed field ablation

SUMMARY:
Various methods exist for performing pulmonary vein isolation (PVI) in patients with atrial fibrillation (AF), including thermal ablation and pulse-field ablation (PFA). However, in cases requiring a second PVI for recurrent AF, radiofrequency ablation (RFA) is utilized in nearly 95% of instances post-acquiring a 3D high-density map from the left atrium (LA). Up to 85% of patients experiencing recurrent AF after the initial PVI exhibit pulmonary vein (PV) reconnections, often identified as the cause of AF.

PFA has demonstrated its safety and efficiency compared to RFA as a swift technique for performing ablation. Yet, whether PFA or RFA stands out as superior or safer when applied for a second PVI remains unclear, as no randomized controlled trial has investigated this comparison. The proposed REPEAT-AF trial aims to randomize 154 AF patients experiencing recurrent AF after the initial PVI, assigning them in a 1:1 ratio to either RFA or PFA. Each patient will receive an implantable cardiac monitor to precisely detect any AF recurrences.

DETAILED DESCRIPTION:
All participating patients are required to provide written (or equivalent) informed consent, indicated by a dated signature of the subject or legal representative. The consent process must comply with applicable national regulations and use language understandable by the patient.

The study will be conducted at 6 clinical centres/investigational sites across the Netherlands. Patients will be randomized (1:1) into a PFA or point-by-point RF ablation arm. Randomization will occur prior to the ablation procedure. A implantable cardiac monitor will be implanted in all randomised patients one month before ablation to accurately monitor any AF/atrial flutter (AFL)/ atrial tachycardia (AT) recurrence. Treatment allocation will be processed through the Dutch 'National Heart Registry' (NHR) data platform.

Patients randomized to both arms of the study will be evaluated for PV isolation at the start of the ablation procedure. If PV reconnection is identified in patients in the point-by-point RF arm, re-ablation will occur according to the study protocol. Patients in the PFA arm will have PV reconnection determined using the FARAWAVE catheter. Those with no PV reconnection (100% PV isolation/durable PVI) will be followed in an observational registry.

The PFA ablation arm involves the use of the Farastar generator system, Farawave ablation catheter, and Faradrive steering catheter for the procedure. The RF point-by-point ablation arm (control) involves RF ablation following standard practice.

ELIGIBILITY:
Subjects who meet all of the following inclusion criteria at screening will be eligible for enrolment:

* Patient had 1 previous PVI with either cryoballoon, RF ablation or PFA
* Index PVI occurred within <5 years prior to enrolment
* Documented AF recurrence >30 seconds
* Symptomatic AF
* Paroxysmal AF
* Age >18 and <80 years
* Willing and capable to provide informed consent
* Able and willing to participate in all examinations and follow-up visits and tests associated with this clinical study

Subjects who meet ANY of the following exclusion criteria will be excluded from the study:

* Persistent AF (by diagnosis of duration >7 days)
* Concomitant/ prior diagnosis for atrial tachycardia (AT) and/or atrial flutter (AFl). Note typical cavotricuspid isthmus dependent flutter is not an exclusion criterium.
* Underwent additional ablations outside the pulmonary veins during index AF ablation
* AF secondary to electrolyte imbalance, thyroid disease, alcohol abuse, or other reversible/non-cardiac causes
* Contraindication to, or unwillingness to use, systematic anticoagulation
* Left ventricular ejection fraction (LVEF) <30% as documented by transthoracic echo (TTE) (within <3 months prior)
* Left atrial volume index >60 ml/m2
* Clinically significant arrhythmias other than AF
* Previous surgery for AF
* New York Heart Association (NYHA) Functional Class III or IV
* Presence of intramural thrombus, tumour or other abnormality that precludes safe catheter introduction or manipulation
* BMI >35 kg/m2
* Significant or symptomatic hypotension, bradycardia, or chronotropic incompetence
* Chronic renal insufficiency of <15 mL/min/1.73 m2 or any history of renal dialysis, or history of renal transplant
* Hemodynamically significant valvular disease
* Presence of patent foramen ovale (PFO) or atrial septal defect (ASD) closure device
* History of abnormal bleeding and/or clotting disorder
* History of rheumatic fever
* Severe lung disease, pulmonary hypertension, or any lung disease. Only if involving abnormal blood gases or significant dyspnoea
* Clinically significant systemic infection or sepsis
* Life expectancy <1 year
* Sensitivity to contrast media not controlled by pre-medication
* Any of the following within the 3 months prior to enrolment:

  * Myocardial infarction
  * Unstable angina
  * Percutaneous coronary intervention
  * Heart failure hospitalization
  * Stroke or TIA
  * Significant bleeding
  * Pericarditis/effusions
  * Left atrial thrombus
* Coronary artery bypass grafting/atriotomy within 6 months prior
* Organ or haematologic transplant, or currently being evaluated for an organ transplant
* Women who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of repeat pulmonary vein isolation (PVI) with PFA or point-by-point RF ablation. | 12 months
  12-month incidence of AF/AFl/AT recurrence.

SECONDARY OUTCOMES:
To compare the efficacy of repeat pulmonary vein isolation (PVI) with PFA or point-by-point RF ablation. | 24 months
  24-month incidence of AF/AFl/AT recurrence.
Repeat PVI within 12 and 24 months of randomization | 12 and 24 months
  Repeat PVI
AF burden with and without 3 months blanking period | 12 and 24 months
  Proportion of cumulative time in AF divided by the total time accrued over follow-up
Change in quality of life | 12 and 24 months
  As measured by EuroQol-5D-5L questionnaire
Change in quality of life as affected by AF | 12 and 24 months
  As measured by AF Effect On Quality-Of-Life (AFEQT) questionnaire
AF hospitalisation / urgent visit | 12 and 24 months
  Hospitalization/urgent visit for atrial fibrillation
Cost-effectiveness | 12 and 24 months
  Cost-effectiveness
Rate of ischemic stroke | 12 and 24 months (efficacy)
  Rate of ischemic stroke
Complications of ablation | 0-30 days post ablation
  Death, stroke, pericarditis, cardiac tamponade, vascular access complications etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Blaauw, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No